CLINICAL TRIAL: NCT06008821
Title: Bilateral Paravertebral Blockade for Improvement of Quality of Recovery Following Cardiac Surgery (P-QOR): a Randomized Controlled Trial
Brief Title: Paravertebral Block for Improvement of Quality of Recovery Following Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Providence Health & Services (Other); Canadian Anesthesiologists' Society (Other)
Responsible Party: Principal Investigator, Terri Sun, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H23-00055
Record Dates: First submitted 2023-07-18; First posted 2023-08-24 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-08

CONDITIONS: Post-operative Pain; Post-cardiac Surgery; Cardiac Disease
Keywords: Regional anesthesia; Paravertebral blockade; Cardiac surgery; Post-operative pain; Quality of recovery
MeSH Terms: conditions — Pain, Postoperative; Heart Diseases | interventions — Epinephrine; Saline Solution

STUDY DESIGN:
Intervention Model Description: This will be a triple-blinded (patient, outcomes assessor and all clinicians except the regional anesthesiologist), individually-randomized, placebo-controlled trial in which patients will be randomly allocated to two study groups in a 1:1 ratio. We will randomize patients in blocks of 4 or 6.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study observes blinding of the patients, anesthesiologists, surgeons, nurses, outcome collectors, and data analysts. Only the regional anesthesiologist performing the intervention will be unblinded. To maintain the quality and legitimacy of the trial, unblinding may only occur if knowledge of the actual intervention is essential to treat and manage the patient. In events such as acute and limited episode of hypotension or bradycardia from a vasovagal event, blinding will be maintained as knowledge of intervention is not required for management. All code breaks with reason will be documented and reported. A protocol description of conditions and procedures for emergency unblinding will be drafted, but the ultimate decision at the time of the block will be at the discretion of the regional anesthesiologist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Bilateral, single level, paravertebral blockade with 0.25% ropivicaine
  Interventions: Procedure: Bilateral paravertebral block with 0.25% ropivicaine with 1:400,000 epinephrine
- Control Group (Sham Comparator): Bilateral, single level, subcutaneous sham block with normal saline
  Interventions: Procedure: Bilateral sham block with normal saline

INTERVENTIONS:
Procedure: Bilateral paravertebral block with 0.25% ropivicaine with 1:400,000 epinephrine — 60mL of 0.25% ropivacaine will be injected into the PVB at thoracic vertebrae T3/4 level bilaterally (30mL at each site for a total of 2 injections)
  Arms: Intervention Group
Procedure: Bilateral sham block with normal saline — 10 mL of normal saline will be injected into subcutaneous space at the T3/4 level bilaterally (5 mL at each site for a total of 2 injections)
  Arms: Control Group

SUMMARY:
This study aims to evaluate the efficacy of bilateral, paravertebral blockade (intervention) against sham blocks (control) placed prior to sternotomy in improving quality of recovery following cardiac surgery.

Primary outcome: The hypothesis is that bilateral single-shot PVB at the thoracic spinal segmental levels T3/4, compared with sham blocks, improve the Quality of Recovery-15 (QoR-15) score at 24 hours following cardiac surgery by a minimally clinically important difference of 8.0 or greater.

Secondary outcomes: The hypothesis is that the intervention will reduce pain scores, opioid requirements, and related side effects; improve respiratory mechanics; and facilitate a better first night's rest/sleep in the first 24-48 hours compared to sham blocks.

DETAILED DESCRIPTION:
This will be a triple-blinded, individually-randomized, single-centered, placebo-controlled trial in which patients will be randomly allocated to two study groups in a 1:1 ratio.

Randomization: The investigators will randomize patients in blocks of 4 or 6. The randomization sequence will be generated online using Sealed Envelope (sealedenvelope.com) . Allocation to treatment versus control will be placed in sealed envelopes. The envelopes will be sequentially numbered, signed and opaque, with the randomization group insert wrapped in foil, and further blocked by carbon paper. On the day of surgery, the regional anesthesiologist be provided the envelope by the research assistant. They will to open it in private, and then destroy its contents immediately upon reading the allocation card.

This study observes blinding of the patients, anesthesiologists, surgeons, nurses, outcome collectors, and data analysts. Only the regional anesthesiologist performing the intervention will be unblinded. To preserve blinding for everyone else, only the regional anesthesiologist and anesthesia assistant will be present in the room at the time of block. Windows on the operating room doors will be covered and a sign mounted to limit entry unless there is an emergency.

Eligible patients will be identified in the Pre-assessment Clinic (PAC) or the inpatient ward. Potentially eligible participants will be screened for significant cognitive impairment, and those scoring 1-2 on the Mini-Cog will be excluded. Enrolled patients will complete a baseline QoR-15 survey. Patients will then be provided a study information package which they can then review on their own time. On the day of surgery, the unblinded regional anesthesiologist will receive information on patient allocation from sealedenvelopes.com and perform the study procedure in the operating room with arterial line monitoring prior to induction of anesthesia. anesthesiologist.

Patients will remain intubated following surgery and be transferred to the CSICU where they are usually extubated within 4-6 hours. Following extubation, patients will receive pain management using hydromorphone IV until transfer to the ward or for the first 24 hours (whichever comes first). For the remainder of the study, the patient will be prescribed a standard postoperative pain control regimen and management will be at the discretion of attending CSICU intensivist, cardiac surgeon or nurse practitioner without influence from this study.

All patients will be followed from the time of randomization thereafter until the common study end date (to be determined, approximately 2 years after the first patient randomized). Primary analysis will be intent to treat.

Statistical Analysis

Sample size: A sample size of n = 112 per group, or total of N=224 patients will be required to reject a null hypothesis that there is no difference in QoR-15 at 24 hours (Student's t test), at a 2-sided alpha of 0.05, and a power of 80% (UBC Sample Size Calculator). This is based off a Minimally Clinically Important Difference of 8.0 in a mixed population of surgical patients reported by Myles et al. At St. Paul's Hospital, the investigators conducted a preliminary prospective study assessing QoR-15 scores in 70 patients approximately 24 hours following cardiac surgery found a lower mean (SD) QoR-15 score of 83.47 +/- 19.86 (unpublished data) than what has been published in the original validation study of QoR-15. The investigators used the QoR-15 scores at 24 hours and a MCID of 8 to calculate a sample size of n=97 per arm. The sample size will be increased by 15% to account for a dropout rate of 5% and delirium rate of 10% observed at St Paul's Hospital, to arrive at a sample size of n=112 per group, or total of N=224 for the entire study.

Primary analysis: intention-to-treat comparison on QoR-15 score at 24 hours (PVB vs sham block) using Student's t test or Mann-Whitney U test). There will be a secondary efficacy analysis done for per protocol population, which would exclude major protocol deviations. In addition, the investigators will conduct a multiple linear regression analysis between the primary outcome of QoR-15 score at 24 hours and treatment group adjusted for baseline QoR-15 score and baseline characteristics (age, sex, history of chronic pain prior to surgery, history depression requiring medication, history of anxiety requiring medication, history of poorly-controlled post-surgical pain, surgical risk stratification (Euroscore II). The primary analyses will be conducted at a two-sided significance level of 0.05

Secondary Analysis: Continuous variables including cumulative opioid consumption, simplified PONVIS score, VISmax score, duration of mechanical ventilation and length of stay will be compared using Student's t test or Mann-Whitney U test, or repeated measures ANOVA with Bonferoni correction when applicable. Dichotomous variables such as atrial fibrillation, pulmonary complications, delirium, and adverse events will be compared using Chi-Squared test or Fisher's Exact Test, or repeated measures ANOVA with Bonferroni correction when applicable. Area under the pain intensity curve (AUE) derived from NRS-11 pain scores obtained from the 4th to 48th hour, and QoR-15 scores at baseline, 24 hours, 48 hours and 12 weeks will be analyzed using a mixed models for repeated measures (MMRM), with baseline values, study group, study visit, and the interaction between study visit and study group as covariates. The analysis of secondary outcomes will be conducted at a two-sided significance level of 0.05.

Handling of Missing data: There will be a proportion of patients who will have missing outcomes due to complications such as delirium/confusion, delayed extubation, postoperative bleeding, and hemodynamic instability. It is anticipated that the loss to follow-up to be <15% which is considered in the sample size calculation. All efforts will be made to collect complete data for all patients in this study. Patients will be followed till the study end and will complete all required data collection. In general, missing values observed in the study will be treated as 'missing'. No attempt will be made to impute missing values and only observed values will be used for analysis.

Subgroup and Sensitivity Analysis: The investigators plan to conduct 3 subgroup analyses based on sex, age, and patients with moderate to severe asthma or COPD. Sensitivity analysis will be conducted comparing intent to treat versus per protocol analysis.

ELIGIBILITY:
Inclusion Criteria

* All adult (19 years or older)
* English-speaking patients
* Scheduled for elective cardiac surgery with full median sternotomy.

Exclusion Criteria

* Patient refusal, inability to provide consent
* Mini-Cog© Score of 1-2
* emergent surgery
* infection at the site of injection
* empyema
* neoplastic mass in the paravertebral space
* known preoperative coagulopathy
* platelet count < 50 x 109, INR or aPTT exceeding the upper range of normal in the absence of anticoagulant use, patients receiving anticoagulation medications or non-ASA anti-platelet medications that have not been stopped for the appropriate duration in accordance with American Society of Regional Anesthesia and Pain Medicine guidelines (20)
* severe kyphoscoliosis or deformed spines or previous thoracic surgery
* allergy to study medications
* preoperative liver failure (as defined by Child-Pugh B or C)
* chronic pain or opioid use history, alcohol or drug use disorders, major psychiatric or neurodevelopmental disorders
* Moderate to severe pain at baseline.
* preoperative renal failure (as defined by eGFR < 30 mL/min/1.73 m2)
* extremes of weight (BMI > 40 kg/m2, and weight < 50 kg)
* Patients anticipated to require prolonged post-operative ventilation > 24 hours after surgery

  * High risk by Euroscore II >=8%) (21-23)
  * 3 or more major procedures
  * Procedures requiring deep hypothermic circulatory arrest (DHCA)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Initial Quality of Recover-15 (QoR-15) score | 24 hours following the intervention
  The QoR-15 score is a validated tool used to assess the quality of recovery at 24 hours. following the intervention. This score ranges from 0 to 150, with higher scores indicating higher quality of recovery.

SECONDARY OUTCOMES:
Subsequent Quality of Recovery-15 (QoR-15) scores | 48 hours following surgery and 12 weeks following surgery
  QoR-15 score at 48 hours following PVB and at 12 weeks following surgery. This score ranges from 0 to 150, with higher scores indicating higher quality of recovery.
Quality of sleep | 24 hours and 48 hours following surgery
  Quality of sleep on the first and second night as measured by Richards-Campbell Sleep Questionnaire. The RCSQ is scored on a visual analogue scale from 0-100, with higher scores representing better sleep.
Opioid consumption | 24 hours and 48 hours following surgery
  Cumulative opioid consumption (in intravenous morphine equivalents) at 24 and 48 hours
Pain scores | every 4 hours for the first 24 hours then every 8 hours until the 48 hour mark following surgery
  Numeric rating scale pain scores at rest and with coughing every 4-8 hours following extubation for 48 hours following the PVB. The bedside nurse will be trained and provided a standardized script to assess pain every 4-8 hours by NRS for the first 48 hours. Pain scores Coughing will be elicited with a standardized script for a sitting patient: "Please use both hands to hold on to the pillow in front you to hold your chest in, and give me three forceful coughs in a row". The pain score ranges from 0-10, with higher score indicating a higher severity of pain.
Severity of post-operative nausea and vomiting | 24 hours and 48 hours following surgery.
  Severity of nausea and vomiting at 24 and 48 hours as measured by the simplified Postoperative Nausea and Vomiting Intensity Scale (PONVIS) using the Impact Score, where clinically significant PONV is defined as having a score of >=5.
Duration of post-operative mechanical ventilation | Up to time of hospital discharge or 14 days post-operatively, whichever is sooner.
  Total duration of post-operative mechanical ventilation will be calculated as the duration of time from arrive in CSICU to first tracheal extubation, up to time of hospital discharge or 14 days post operatively, which ever is sooner. Extubation time will be obtained from respiratory therapy notes.
Incidence of pulmonary complications | 24 hours and 48 hours following surgery
  Pulmonary complications at the 24 and 48 hr mark will be recorded by the research assistant after consulting with the nurse and or physician in charge. Pulmonary complications will include respiratory events requiring defined as non-invasive positive pressure ventilation or high flow nasal cannula or non-rebreather mask, tracheal reintubation, >5L NP or face mask oxygenation. It will be assessed from date of randomization up to 48 hours following surgery.
Incidence of new onset post-operative atrial fibrillation | Up to 48 hours following surgery
  New onset post operative atrial fibrillation (defined as persistent or ≥2 paroxysmal episodes lasting >24 hours) will be collected at the time of hospital discharge. It will be assessed from date of randomization until the date of first documented occurrence assessed up to 48 hours following surgery.
Incidence of new onset delirium during hospital stay | Up to time of hospital discharge or 14 days post-operatively, whichever is sooner.
  Delirium as per CAM-ICU will be reviewed and noted as "present" or "absent" . It will be assessed from date of randomization until the date of first documented occurrence assessed up to hospital discharge or 14 days post-operatively, whichever is sooner.
Incidence of hospital or ventilator acquired pneumonia during hospital stay | Up to time of hospital discharge or 14 days post-operatively, whichever is sooner.
  Hospital or ventilator acquired pneumonia requiring antibiotics will be reviewed after discharge from discharge summary. It will be assessed from date of randomization until the date of first documented occurrence assessed up to hospital discharge, or 14 days postoperatively, whichever is sooner.
Cardiac Surgery Intensive Care unit length of stay | Up to time of hospital discharge or 14 days post-operatively, whichever is sooner.
  CSICU length of stay (days) will be defined from time of arrival to CSICU post operatively to time that the patient is ready (but not necessarily physically transferred) for the ward, as determined by nursing. It will be collected by bedside nursing prior the patient leaving the cardiac surgery intensive care unit.
Hospital length of stay | Up to time of hospital discharge or 14 days post-operatively, whichever is sooner.
  Duration of hospital length of stay (days) will be collected at the time of discharge, or 14 days post-operatively, whichever is sooner.

CONTACTS AND LOCATIONS:
Overall Officials: Terri Sun, M.D., Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No